CLINICAL TRIAL: NCT01013194
Title: Human Fetal Liver Cell Transplantation for Treatment of Chronic Liver Failure
Brief Title: Human Fetal Liver Cell Transplantation in Chronic Liver Failure
Acronym: hFLCTx
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRRB/01/06
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; Fetal stem cells; Stem cell transplantation; Liver transplant candidate
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated patients (Experimental): Cirrhotic patients treated with Human Fetal Liver Cell Transplantation.
  Interventions: Other: Human Fetal Liver Cell Transplantation
- Control patients (No Intervention): Cirrhotic patients on Standard therapy.

INTERVENTIONS:
Other: Human Fetal Liver Cell Transplantation — Human Fetal Liver Cell Transplantation. Cell source: Non-purified and non-selected fetal liver cells from fetuses aborted between the 16th and 26th week of gestation.
  Infusion technique: Isolation and incannulation of the femoral artery.Splenic artery infusion under radiological guidance.
  Cell infusion: between 5 and 10x10^8 cells. Number of sessions: up to 2.
  Arms: Treated patients

SUMMARY:
The herein study consists in the transplantation of liver progenitor cells isolated from human fetal liver tissue with the aim of improving conventional liver therapy and broadening therapeutical options other than liver transplantation.

DETAILED DESCRIPTION:
One of the major clinical problems in transplantation medicine is the discrepancy between the growing number of liver chronic disease patients and the lack of organs. Research and development of new liver failure treatments thus have a high clinical significance. Regenerative medicine and results recently achieved in the field of stem cell biology may provide a remedy to this emerging problem.

Our project aims at developing new generation cell transplantation methodologies through an interdisciplinary research project created from a collaboration between ISMETT, Palermo and the University of Pittsburgh (UPMC-USA).

Adult hepatocyte transplantation has been in use for several years already and has proved to be safe for patients and able, especially in pediatric patients, to improve liver function indices and delay the need for liver transplantation. Studies have been limited until now by the use of already differentiated hepatocytes and therefore unable to proliferate and develop a suitable liver mass to support a decompensated liver.

The hypothesis of our project, supported by in vitro studies and studies on experimental animal models, is based on the possibility to generate an ectopic liver system in the spleen through the experimental use of hepatic cell progenitors obtained from human fetal liver tissues. Human fetal liver cell transplantation will be performed in the spleen through arterial injection.

The final endpoint of the project is to develop an innovative and safe treatment for patients with end-stage chronic liver failure

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis (evidence of chronic liver disease, presence of ascites and/or esophageal varices upon superior digestive endoscopy and/or ultrasound evidence of portal hypertension) or histological diagnosis of liver cirrhosis with any etiology.
* Serious liver failure documented by a score ≥ B8 based on the Child-Pugh-Turcotte classification and/or MELD score ≥ 14.
* Informed consent to the study signed by the patient.

Exclusion Criteria:

* MELD score ≥ 25
* Hepatocellular carcinoma (HCC)
* Portal vein thrombosis
* Serious cardiovascular or respiratory disease, or other medical condition which may threaten patient's life in the subsequent three months
* Admission to the Intensive Care Unit (ICU)
* Hemodynamic instability (MAP < 55 mmHg)
* Use of vasoactive drugs (Epinephrine, Norepinephrine, Vasopressin, Dopamine, Terlipressine
* Type-1 (acute) hepatorenal syndrome
* Levels of serum creatinine >2 mg/dl and/or creatinine clearance <30-40 ml/min
* Sepsis, active infection or spontaneous bacterial peritonitis
* Active gastrointestinal bleeding or recent gastrointestinal bleeding episode (in the previous 4 weeks)
* Active alcohol abuse
* Severe alcoholic hepatitis
* Pulmonary hypertension (PAP > 35 mmHg)
* History of neoplasia
* Pregnancy
* Non Sicilian residency
* HBV DNA positive
* HIV infection
* Drug addiction
* Age < 18 years
* Transjugular intrahepatic portosystemic shunt (TIPS) placed in the previous month
* Contraindications to the procedure (e.g., related to the splenic artery: aneurysm, kinking, thrombosis, splenic-renal shunt; related to the spleen: large angioma).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gridelli, MD, Principal Investigator — ISMETT-UPMC
Locations (1):
- ISMETT, Palermo, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Patients: Cell source: Non-purified and non-selected fetal liver cells from fetuses aborted between the 16th and 26th week of gestation.
  Infusion technique: Isolation and incannulation of the femoral artery.Splenic artery infusion under radiological guidance.
  Cell infusion: between 5x10^8 and 10x10^8 cells. Number of sessions: up to 2.
- Control Group: Cirrhotic patients in waiting list for Liver Transplantation on standard therapy
Period: Overall Study
Arm/Group | Treated Patients | Control Group
Started | 9 | 16
Completed | 9 (Consecutive patients) | 16 (Retrospectively contemporary matched-pair group)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treated Patients: Patients with end-stage chronic liver disease in waiting list for liver transplantation treated with non-purified and non-selected fetal liver cells.
- Control Patients: Patients with end-stage chronic liver disease on standard therapy in waiting list for liver transplantation.
- Total: Total of all reporting groups
Arm/Group | Treated Patients | Control Patients | Total
Number analyzed (Participants) | 9 | 16 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 16 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  Italy | 9 | 16 | 25

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival
Description: Assessment of treated and control patients survival at 1 year follow-up
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Treated Patients: Patients with end-stage chronic liver disease in waiting list for Liver Transplantation treated with hFLCTx
- Control Patients: Patients with end-stage chronic liver disease in waiting list for Liver Transplantation on standard therapy
Arm/Group | Treated Patients | Control Patients
Number analyzed (Participants) | 9 | 16
participants
  Patient survival | 5 | 6
  Death/Transplant | 4 | 10
Statistical Analysis 1: Comparison: Treated Patients vs Control Patients; Test type: Superiority or Other; p = 0.4340, Fisher Exact

2. Secondary Outcome: Analysis of Child-Pugh Score From Baseline to 1 Year Follow-up
Description: Assessment of the efficacy of human fetal liver progenitor cell transplantation on Child-Pugh score.
  The Child-Pugh (CP) classification is a scoring system used for the classification of the severity of cirrhosis. It includes three continuous variables (bilirubin, albumin and INR) and two discrete variables (ascites and encephalopathy). Each variable is scored 1-3 with 3 indicating most severe derangement. The determination of CP score may range from 5 to 15 and the final score allows to categorize patients in Child-Pugh A (5-6 points), B (7-9 points) and C (10-15 points). The highest is the score the sickest is the patient.
Time Frame: Baseline and 1 year Follow-up
Population: Baseline Child-Pugh score vs Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treated Patients: Cirrhotic patients in waiting list for Liver Transplantation treated with non-purified and non-selected fetal liver stem cells
Arm/Group | Treated Patients | Control Group
Number analyzed (Participants) | 9 | 16
units on a scale
  Baseline Child-Pugh score | 10.11 (1.54) | 10.00 (1.26)
  Follow-up Child-Pugh score | 9.11 (1.45) | 11.13 (1.63)
Statistical Analysis 1: Comparison: Treated Patients vs Control Group; Comparison at 1 year Follow-up; Test type: Superiority or Other; p = 0.0076, t-test, 2 sided

3. Secondary Outcome: Analysis of Meld Score From Baseline to 1 Year Follow-up
Description: Assessment of the efficacy of human fetal liver progenitor cell transplantation on Meld score.
  The Model for End-stage Liver Disease (MELD) scoring system aims at stratifying recipients by their disease severity according to a score estimating the 3-month probability of death on the waiting list. The calculation of an individual's MELD score is based on three objective lab parameters (bilirubin, serum creatinine and prothrombin time expressed as international normalized ratio, INR) and it includes logarithmic transformations and multiplication by several factors. It ranges between 6 and 40. The highest is the score the lower is the patient's survival.
Time Frame: Baseline and 1 year Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Patients: Cirrhotic patients in waiting list for Liver Transplantation on standard therapy
Arm/Group | Treated Patients | Control Patients
Number analyzed (Participants) | 9 | 16
units on a scale
  Baseline Meld score | 16.00 (2.96) | 15.31 (2.50)
  Follow-up Meld score | 15.67 (3.84) | 19.06 (5.70)
Statistical Analysis 1: Comparison: Treated Patients vs Control Patients; Comparison at 1 year Follow-up; Test type: Superiority or Other; p = 0.0437, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Treated Patients: Patients with end-stage chronic liver disease in waiting list for liver transplantation treated with non-purified and non-selected fetal liver cells from fetuses aborted between the 16th and 26th week of gestation.
- Control Group: Patients with end-stage chronic liver disease in waiting list for liver transplantation.
Arm/Group | Treated Patients | Control Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/16
Other Adverse Events (participants affected / at risk) | 0/9 | 0/16

LIMITATIONS AND CAVEATS:
Using a single gynecology unit we had only a 22% rate of fetal donation, necessarily limiting the availability of hFLCs. Our strict inclusion criteria limited the pool of potential patients to enroll.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes